CLINICAL TRIAL: NCT06245174
Title: NeuroVision™: A Smartphone Application for Neurology and Telemedicine
Brief Title: A Smartphone Application for Neurology and Telemedicine
Acronym: NeuroVision
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Altec Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: R43NS125709 (NIH); R43NS125709 (NIH)
Record Dates: First submitted 2024-01-15; First posted 2024-02-07 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease(PD)
Keywords: Movement Disorders; Parkinson's Disease; 3D Camera; Smartphone; Motor Assessment; Telehealth
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease (PD): Individuals with mild to severe movement disorder symptoms of Parkinson's disease

SUMMARY:
This observational research study is designed to assess the feasibility of developing a new software application that can be used in the home using a commercially available camera to measure abnormal body movements associated with Parkinson's disease (PD). The goal of this study is to validate the motor outcomes derived from a consumer camera observing a sub-set of standardized assessment tasks with respect to the reference motion capture system.

DETAILED DESCRIPTION:
The long-term goal of this project is to develop a new software application (NeuroVision App) for a smartphone or tablet that can be used in the home to measure abnormal body movements associated with Parkinson's disease (PD). The outcomes are intended to enhance PD symptom monitoring in the context of telehealth videoconferences with a clinician. Typical abnormal body movements that can be assessed with the proposed solution include uncontrolled shaking of hands and limbs (tremor) or spastic movements (dyskinesia) while at rest; abnormally slow movements when reaching or walking (bradykinesia); or inability to initiate a movement (akinesia) using 5 standardized motor assessment tasks (sitting at rest, walking, finger tapping, foot tapping, and foot stomping) derived from the Unified Parkinsons Disease Rating Scale (UPDRS). The proposed solution will make it easier for the doctor to periodically assess the motor signs of PD during remote telehealth appointments which may be more convenient and safer for the patient. Current reliance on videoconferencing apps make it difficult to record and measure such symptoms accurately in a telehealth setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female;
* 35 years of age or older;
* Physician-diagnosed Parkinson's disease or other movement disorder such as Essential Tremor or Dystonia;
* One or more mild to moderate motor symptoms of PD (tremor, bradykinesia, akinesia, Parkinsonian gait);
* Hohn and Yahr (Stage I-III);
* Independent ambulator - walker or cane allowed;
* Referring neurologist indicates that prospective subject is not at high fall risk and can safely participate in the study;
* Have participated in prior telehealth visits using videoconferencing app;
* Have used a smartphone in past to record videos;
* Able to provide his/her written informed consent to participate in the study as stated in the informed consent document;
* American-English speaking; able to follow directions in English;
* Normal hearing.

Exclusion Criteria:

* Inability to understand spoken English or follow simple instructions;
* Inability to provide written informed consent.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons who have Parkinson's disease under a doctor's care for movement disorder management at a primary-care or specialty (neurology) out-patient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Tremor Duration | 2 minute
  Duration in seconds of resting tremor in the hands obtained using the NeuroVision prototype while the subject is sitting at rest.
Tremor Amplitude | 2 minute
  Amplitude in centimeters of resting tremor in the hands obtained using the NeuroVision prototype while the subject is sitting at rest.
Parkinsonian Gait - Step Length | 5 minute
  Step length in centimeters obtained using the NeuroVision prototype while the subject is walking.
Parkinsonian Gait - Step Time | 5 minute
  Step time in seconds obtained using the NeuroVision prototype while the subject is walking.
Parkinsonian Gait - Step Variability | 5 minute
  Step variability in centimeters obtained using the NeuroVision prototype while the subject is walking.
Bradykinesia Finger Tap Duration | 2 minute
  Duration in seconds of a finger tapping task obtained using the NeuroVision prototype while the subject opens and closes their hand as rapidly as possible.
Bradykinesia Finger Tap Amplitude | 2 minute
  Amplitude in centimeters of a finger tapping task obtained using the NeuroVision prototype while the subject opens and closes their hand as rapidly as possible.
Bradykinesia Foot Tap Duration | 2 minute
  Duration in seconds of a foot tapping task obtained using the NeuroVision prototype while the subject taps their toes on the floor as rapidly as possible.
Bradykinesia Foot Tap Amplitude | 2 minute
  Amplitude in centimeters of a foot tapping task obtained using the NeuroVision prototype while the subject taps their toes on the floor as rapidly as possible.
Bradykinesia Foot Stomping Duration | 2 minute
  Duration in seconds of a foot stomping task obtained using the NeuroVision prototype while the subject lifts and lowers their foot on the floor as rapidly as possible.
Bradykinesia Foot Stomping Amplitude | 2 minute
  Amplitude in centimeters of a foot stomping task obtained using the NeuroVision prototype while the subject lifts and lowers their foot on the floor as rapidly as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Bhawna Shiwani, MS, Principal Investigator — Senior Research Scientist
Locations (1):
- Altec Inc., Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No